CLINICAL TRIAL: NCT03028298
Title: Sildenafil for the Treatment of Delayed Cerebral Ischemia Following Subarachnoid Hemorrhage
Brief Title: Sildenafil for DCI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0134
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Vasospasm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either low dose sildenafil (20mg oral and 10mg intravenous) or high dose sildenafil (60mg oral and 30 mg intravenous)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose sildenafil (Experimental): Twelve patients with cerebral vasospasm following aneurysmal subarachnoid hemorrhage will be assigned to low dose sildenafil citrate and will receive a 20mg oral dose and a subsequent 10mg intravenous dose of sildenafil citrate.
  Interventions: Drug: Low dose sildenafil citrate
- High dose sildenafil (Experimental): Twelve patients with cerebral vasospasm following aneurysmal subarachnoid hemorrhage will be assigned to high dose sildenafil citrate and will receive a 60mg oral dose and a subsequent 30mg intravenous dose of sildenafil citrate.
  Interventions: Drug: High dose sildenafil citrate

INTERVENTIONS:
Drug: Low dose sildenafil citrate
  Arms: Low dose sildenafil
Drug: High dose sildenafil citrate
  Arms: High dose sildenafil

SUMMARY:
Each year, approximately 30,000 people in the United States suffer an intra-cranial hemorrhage due to aneurysmal rupture. Of those surviving the initial event, up to 40% will go on to have further neurological injury secondary to stroke (delayed cerebral ischemia) caused by constriction of blood vessels (i.e. vasospasm). Previous studies have shown that the medication sildenafil, given intravenously, improves vasospasm, but has an associated degree of hypotension. The degree of hypotension was well within safety thresholds for these patients.

Sildenafil is a medication that strongly inhibits the protein phosphodiesterase-V (PDE-V). The hypothesis for this study is that oral sildenafil will also improve vasospasm, but does not result in as much hypotension. Specifically, the investigators look to show that comparable doses of oral sildenafil produces the same degree of PDE-V inhibition as an intravenous dose while the degree of hypotension is reduced. Additionally, using measurements of cerebral blood flow regulation acquired using transcranial Doppler ultrasound, the investigators look to show that oral sildenafil produces the same degree of improvement in vasospasm and blood flow regulation.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 21
2. Onset of symptoms within 72 hours from presentation
3. Subarachnoid hemorrhage from ruptured cerebral aneurysm
4. Cerebral vasospasm diagnosed on transcranial doppler, CT angiography, or digital subtraction angiography

Exclusion Criteria:

1. Pregnancy
2. Subarachnoid hemorrhage secondary to traumatic or mycotic aneurysm
3. Pre-ictal sildenafil therapy (last dose within 1 week of presentation)
4. Contraindications to sildenafil therapy (i.e. use of nitrates, left ventricular outflow obstruction, impaired autonomic blood pressure control)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-12; Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean arterial blood pressure | baseline and 2 hours post-dose
Area under the plasma concentration versus time curve (AUC) of sildenafil | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 16, 20, and 24 hours post-dose

SECONDARY OUTCOMES:
Area under the cerebral spinal fluid concentration versus time curve (AUC) of sildenafil | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 16, 20, and 24 hours post-dose
Change from baseline in cerebral autoregulation | baseline and 2 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Chad W Washington, MS, MD, MPHS, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Washington CW, Derdeyn CP, Dhar R, Arias EJ, Chicoine MR, Cross DT, Dacey RG Jr, Han BH, Moran CJ, Rich KM, Vellimana AK, Zipfel GJ. A Phase I proof-of-concept and safety trial of sildenafil to treat cerebral vasospasm following subarachnoid hemorrhage. J Neurosurg. 2016 Feb;124(2):318-27. doi: 10.3171/2015.2.JNS142752. Epub 2015 Aug 28. PMID 26314998
- [Background] Dhar R, Washington C, Diringer M, Zazulia A, Jafri H, Derdeyn C, Zipfel G. Acute Effect of Intravenous Sildenafil on Cerebral Blood Flow in Patients with Vasospasm After Subarachnoid Hemorrhage. Neurocrit Care. 2016 Oct;25(2):201-4. doi: 10.1007/s12028-016-0243-0. PMID 26940913